CLINICAL TRIAL: NCT00001281
Title: Studies of the Pathogenesis of HIV Infection in Human Peripheral Blood Cells and/or Body Fluids in People Living With and Without HIV
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910140; 91-I-0140
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-06

CONDITIONS: HIV; Immunodeficiencies; Infectious Diseases
Keywords: Lymphocytes; Venipuncture; Mononuclear Cells; Natural History
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals living with/without HIV: Individuals living with/without HIV
- Individuals living with/without infectious diseases: Individuals living with/without infectious diseases of interest
- Individuals with/without Immunodeficiencies: Individuals with/without immunodeficiencies

SUMMARY:
We are studying virologic and/or immunologic parameters of HIV infection and other infectious or non-infectious immune deficiency diseases in order to better understand the pathogenesis of HIV. Because of the lack of an adequate animal model it is generally necessary to utilize human peripheral blood cells for studying aspects of either in vivo or in vitro HIV infection. We wish to be able to continue to elucidate many pathogenic aspects of HIV infection in relation to other infectious or non-infectious immune regulation and dysregulation using human peripheral blood mononuclear cells as a model....

DETAILED DESCRIPTION:
We are studying virologic and/or immunologic parameters of HIV infection and other infectious or non-infectious immune deficiency diseases in order to better understand the pathogenesis of HIV. Because of the lack of an adequate animal model it is generally necessary to utilize human peripheral blood cells for studying aspects of either in vivo or in vitro HIV infection. We wish to be able to continue to elucidate many pathogenic aspects of HIV infection in relation to other infectious or non-infectious immune regulation and dysregulation using human peripheral blood mononuclear cells as a model.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18 years of age or older.
* Adequate venous access.
* Have a blood pressure less than or equal to 180/100: pulse rate 50-100, unless a lower pulse rate is considered normal for the volunteer.
* Have adequate blood counts (volunteers living with HIV: hemoglobin greater than or equal to 9.0 g/dL, platelets greater than or equal to 50,000; volunteers living without HIV: hemoglobin greater than or equal to 9.0 g/dL, platelets greater than or equal to 50,000
* Be willing and able to provide written informed consent on screening, comply with study requirements and procedures, and comply with clinic policies
* Willingness to allow blood samples to be used for future studies of HIV infection/pathogenesis, and undergo hepatitis screening

EXCLUSION CRITERIA:

* Pregnant and/or breastfeeding females.
* Active substance abuse or history of prior substance abuse that may interfere with protocol compliance or compromise volunteer safety.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers living with/without HIV, Volunteers with/without immunodeficiencies, Volunteers with/without infectious diseases of interest
Sampling Method: Non-Probability Sample
Enrollment: 2419 (Estimated)
Dates: Start 1993-03-09 (Actual)

PRIMARY OUTCOMES:
The purpose of this protocol is to provide a mechanism to obtain blood products and other biologic samples that will be used by NIH Intramural Investigators in studies of HIV and other infectious or immune deficiency diseases | Throughout
  To provide a mechanism to obtain blood products and other biologic samples that will be used by NIH Intramural Investigators in studies of HIV and other infectious or immune deficiency diseases.

SECONDARY OUTCOMES:
To provide the opportunity to compare genomic and proteomic properties of specimens obtained from individuals living with HIV, other infectious diseases, and other immunodeficiencies with those of healthy volunteers | Throughout
  To provide the opportunity to compare genomic and proteomic properties of specimens obtained from individuals living with HIV, other infectious diseases, and other immunodeficiencies with those of healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Moir, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Identified data in BTRIS (automatic for activities in the Clinical Center).@@@@@@@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements.@@@@@@@@@@@@This study will comply with the NIH Genomic Data Sharing Policy, which applies to all NIH-funded research that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data. De-identified data may be shared in an NIH-funded or approved public repositories, including the Database of Genotypes and Phenotypes (dbGAP) or in NCBI Virus Portal for viral sequencing.
Supporting Information: Study Protocol
Time Frame: Shared scientific data should be made accessible as soon as possible, and no later than the time of an associated publication, or the end of the award/support period, whichever comes first.@@@@@@@@@@@@Genomic data will be shared following the guidelines of the Genomic Data Sharing Policy, when applicable.
Access Criteria: Identified data in BTRIS (automatic for activities in the Clinical Center and will be available for use following the BTRIS Policy for Data Sharing and Use).@@@@@@@@@@@@De-identified or identified data with approved outside collaborators under appropriate agreements.@@@@@@@@@@@@De-identified genomic data may be shared in an NIH-funded or approved public repositories, including the Database of Genotypes and Phenotypes (dbGAP) or in NCBI Virus Portal for viral sequencing and the use of the data within will be governed by their policies.

REFERENCES:
- [Background] Jelicic K, Cimbro R, Nawaz F, Huang da W, Zheng X, Yang J, Lempicki RA, Pascuccio M, Van Ryk D, Schwing C, Hiatt J, Okwara N, Wei D, Roby G, David A, Hwang IY, Kehrl JH, Arthos J, Cicala C, Fauci AS. The HIV-1 envelope protein gp120 impairs B cell proliferation by inducing TGF-beta1 production and FcRL4 expression. Nat Immunol. 2013 Dec;14(12):1256-65. doi: 10.1038/ni.2746. Epub 2013 Oct 27. PMID 24162774
- [Background] Le Saout C, Hasley RB, Imamichi H, Tcheung L, Hu Z, Luckey MA, Park JH, Durum SK, Smith M, Rupert AW, Sneller MC, Lane HC, Catalfamo M. Chronic exposure to type-I IFN under lymphopenic conditions alters CD4 T cell homeostasis. PLoS Pathog. 2014 Mar 6;10(3):e1003976. doi: 10.1371/journal.ppat.1003976. eCollection 2014 Mar. PMID 24603698
- [Background] Auerbach DJ, Lin Y, Miao H, Cimbro R, Difiore MJ, Gianolini ME, Furci L, Biswas P, Fauci AS, Lusso P. Identification of the platelet-derived chemokine CXCL4/PF-4 as a broad-spectrum HIV-1 inhibitor. Proc Natl Acad Sci U S A. 2012 Jun 12;109(24):9569-74. doi: 10.1073/pnas.1207314109. Epub 2012 May 29. PMID 22645343
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1991-I-0140.html